CLINICAL TRIAL: NCT04736680
Title: Pediatric Virtual Visits as a Strategy for Access to Care During the COVID-19 Pandemic in a Pediatric Hospital. Missed Appointments Rates, Associated Factors, Generation and Validation of Predictive Models
Brief Title: Pediatric Virtual Visits as a Strategy for Access to Care During the COVID-19 Pandemic in a Pediatric Hospital
Status: Completed | Type: Observational
Sponsor: Hospital General de Niños Pedro de Elizalde (Other)
Responsible Party: Sponsor
Other Study IDs: 2392
Record Dates: First submitted 2021-02-01; First posted 2021-02-03 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Telehealth
Keywords: Telehealth; Children; COVID-19; virtual visit; Lost appointments
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lost Virtual Visit: Pediatric patients who had scheduled an appointment for a virtual visit and missed.
- Attended Virtual Visit: Pediatric patients who had scheduled an appointment for a virtual visit and attended.

SUMMARY:
In this study we will describe the factors associated with missed virtual visit appointments in an academic children´s hospital during the covid-19 pandemic and we will develop a predictive model that serves as the basis for improving the Telehealth Program.

DETAILED DESCRIPTION:
Pediatric visits are a fundamental axis of health policies because actions to promote and protect health have a maximum effect on children. Due to the COVID-19 pandemic a marked decrease in pediatric visits was observed in scheduled and on-call visits. This fact can be explained by the restriction on people's circulation necessary to contain COVID-19 dissemination. In this context, the population that attends the Hospital General de Niños Pedro de Elizalde was especially affected, since 91% of the patients attending the institution live in another district.

In order to overcome this barrier in access to care, we decided to implement a Telehealth Program that uses virtual visits as a tool for access to care. Little is known about the effects that these programs can have on patients with exclusive public health coverage. Although virtual visits could be a solution for access to care in an oversaturated system, there is the possibility that virtual visits could not be carried out and that a significant proportion will be lost, increasing inequity and difficulties in access to health.

Due to the relevance of the topic and the little information available, we propose in this study to estimate the proportion of virtual visits appointments lost. On the other hand, considering the possibility of avoiding the loss of virtual visits appointments, we propose to describe the factors associated with missed appointments and develop a predictive model that serves as the basis for improving the Telehealth Program.

ELIGIBILITY:
Inclusion Criteria:

* All scheduled virtual visits

Exclusion Criteria:

* On-call virtual visits

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All scheduled virtual visit appointments between August 1 2020 and 31 december 2020 will be included. The sample will be randomized to allocate a generation cohort (two-thirds of the sample) and a validation cohort (one third of the sample).
Sampling Method: Non-Probability Sample
Enrollment: 3339 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of missed appointments | 6 months
  Characterize, describe and compare the clinical and administrative characteristics of outpatients who didn't attend and attended an appointment in pediatrics

SECONDARY OUTCOMES:
Clinical and administrative characteristics | 6 months
  Characterize, describe and compare the clinical and administrative characteristics of outpatients who didn't attend and attended an appointment in pediatrics

CONTACTS AND LOCATIONS:
Overall Officials: Mariano E Ibarra, MD, Principal Investigator — Hospital General de Niños Pedro de Elizalde
Locations (1):
- Hospital General de Niños Pedro de Elizalde, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No